CLINICAL TRIAL: NCT01181115
Title: An Open-Label Study to Evaluate the Safety and Tolerability and to Explore the Efficacy of Avonex (Interferon Beta-1a) in Chinese Subjects With Relapsing Multiple Sclerosis
Brief Title: Avonex Safety and Tolerability in Chinese Subjects With Relapsing Multiple Sclerosis (MS)
Acronym: Avonex China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108MS301
Record Dates: First submitted 2010-08-05; First posted 2010-08-13 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Sclerosis
Keywords: Chinese Patients; Relapsing MS; Safety; Avonex; Tolerability; Gadolinium; Interferon Beta 1a
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (Experimental): Interferon treatment for MS
  Interventions: Drug: Avonex

INTERVENTIONS:
Drug: Avonex — Interferon treatment for MS

SUMMARY:
The study is designed to determine the effect of weekly intramuscular (IM) administration of 30 mcg Avonex (interferon beta 1a) on safety parameters and gadolinium (Gd) enhanced and T2-weighted cranial magnetic resonance imaging (MRI) lesions in Chinese patients with clinically diagnosed (using revised McDonald criteria) relapsing multiple sclerosis (MS).

DETAILED DESCRIPTION:
This is a multicenter, open-label, safety study to support registration of Avonex in China by providing data on the effect of weekly IM administration of 30mcg Avonex on safety parameters in Chinese patients with clinically diagnosed relapsing MS. This study will also include an intra-subject exploratory comparison of pre-treatment MRI (at -3 months and at month 0) and post -treatment MRI (at month 3 and month 6). Up to 60 subjects with relapsing forms of MS will be recruited to approximately 6 sites in China.

The study period will consist of screening, a 6 month open-label treatment period, and follow up at 30 days post-dosing. There will be a total of 8 clinic visits and 1 telephone contact.

Screening: will be determined 3 months +/- 7 days prior to subjects' first dose of Avonex on Day 1, at which time a screening MRI with and without Gd-enhancement will be performed.

Treatment Period: consists of eligible patients undergoing pre-dosing assessments and receiving the first dose of Avonex on day 1. Subjects will have a brain MRI within 48 hours prior to the first injection of Avonex.

Weekly doses of open-label Avonex 30mcg IM will be administered for 24 consecutive weeks for a total of 25 injections per subject. Subjects or their caregivers will be allowed to self-inject after successful completion of appropriate IM injection training.

Subjects will return to the clinic at weeks 6, 12, 18 and 24 for safety and laboratory assessments (including blood sample collection for pharmacodynamic (neopterin) and immunogenicity testing), and clinician injection site assessments. Subjects will undergo brain MRI with and without Gd enhancement at week 12 and week 24. Subjects will perform injection site pain assessments on day 1 and at weeks 6, 12, 18, and 24 recording results on a visual analog scale. Subjects who prematurely discontinue Avonex may remain in the study and continue protocol-scheduled visits/evaluations (with the exception of subject and clinician injection site assessments and neopterin sample collection.

Subjects who experience new or worsening symptoms suggestive of an MS relapse will have a neurological worsening visit within 5 days following onset of symptoms. Treatment of confirmed MS relapses will follow a protocol-specified regimen.

Post treatment period: subjects will undergo follow-up assessment at week 24 (at 24+/- 8 hours following their last Avonex injection, if applicable). Subjects will have a telephone follow up contact conducted 30 (+/- 7 days) after their last study visit to assess AEs and use of concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand risks of study and provide informed consent.
* Must be Chinese, aged 18 to 55 years inclusive at time of consent.
* Must have diagnosis of relapsing MS of 3 months duration at time of screening visit.
* Must have at least 1 documented MS attack within 3 years of Day 1.
* Must have EDSS score of 0 to 5 inclusive at screening visit.
* All male subjects & female subjects of child-bearing potential must practice effective contraception during the study.

Exclusion Criteria:

* Have a diagnosis of primary progressive, secondary progressive, or progressive relapsing MS.
* Have had a clinical MS attack within the 50 days prior to Day 1, and or the subject has not stabilized from a previous attack in the opinion of the Investigator.
* The subject is unable to undergo a brain MRI scan for any reason.
* The subject's screening and Day 1 MRIs are both normal (negative) for lesions consistent with MS (Gd-enhancing lesions are not required, but one of the 2 MRIs should be consistent with MS).
* History of severe allergic or anaphylactic reactions.
* Known allergy to any component of the Avonex Formulation.
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal or other major disease.
* Subjects with a history of malignant disease, including solid tumors, and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and considered cured).
* History of seizure disorder or unexplained blackouts OR history of a seizure within 6 months prior to Day 1.
* History of suicidal ideation or an episode of clinically severe depression (as determined by the Investigator) within 6 months prior to Day 1. Note: subjects receiving ongoing antidepressant therapy will not be excluded from the study unless the medication has been increased within the 6 months prior to Day 1.
* Clinically significant abnormal ECG values as determined by the Investigator.
* Known history of human immunodeficiency virus (HIV).
* Known history of, or positive test result for hepatitis C virus (test for hepatitis C virus antibody HCV Ab) or hepatitis B virus (test for Hepatitis B surface Antigen HBsAg) and/or Hepatitis B Core Antibody (HBcAb).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The number and proportion of subjects with adverse events (AEs) | 24 weeks
Assessment of clinical laboratory parameters | 24 weeks
Assessment of vital signs and physical examinations | 24 weeks
Assessment of electrocardiogram (ECG) | 24 weeks
Assessment of immunogenicity | 24 weeks
Incidence of depression | 24 weeks
Incidence of flu-like symptoms | 24 weeks
Subject assessment of injection site pain | 24 weeks
Clinical assessment of the injection site | 24 weeks

SECONDARY OUTCOMES:
Assess safety of Avonex by evaluating changes in the Expanded Disability Status Scale (EDSS) score over time | 24 weeks
Number of Gd-enhancing lesions on brain MRI scans taken after 3 and 6 months following Avonex treatment | at month 3 and month 6
Number of new or newly enlarging T2-weighted lesions on brain MRI scans taken after 3 and 6 months following Avonex treatment | at month 3 and month 6
Volume of T2-weighted lesions on brain MRI scans taken after 6 months following initiation of Avonex treatment | month 6
Assess pharmacodynamic response to Avonex by evaluating the change from baseline in serum levels of neopterin | 24 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Taiyuan
  - Research Site, Xi'an